CLINICAL TRIAL: NCT01702142
Title: To Test a Payer/Treatment Agency Intervention to Increase Use of Buprenorphine
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: Molfenter_2012_0008; 1R01DA030431-01A1 (NIH)
Record Dates: First submitted 2012-09-28; First posted 2012-10-05 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Addiction
Keywords: Addiction Treatment
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Biospecimens are not part of this study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- NIATx Only: NIATx (Network for the Improvement of Addiction Treatment) organization change model only
- NIATx and Advancing Recovery: Organizational and system changes

SUMMARY:
A team of researchers from the University of Wisconsin-Madison College of Engineering and Oregon Health & Science University will test whether clinician training and the use of organizational change strategies are sufficient for disseminating an evidence-based practice (EBP), or if changes to both organizational systems and payer policy results in greater EBP use. Demonstrating the role of payment policy as a driver in the adoption of evidence-based practices could provide a contribution to dissemination and implementation science. This study will employ an intervention that was developed through the Robert Wood Johnson Foundation-funded Advancing Recovery (AR) program. In AR, payer/treatment organization partnerships in 12 states collaborated to remove systemic barriers to the adoption of EBPs such as medication-assisted treatment for substance abuse disorders. The resulting "AR Framework" of payer and organizational change strategies will be tested against its ability to increase the use of the addiction medication buprenorphine as compared to organizational change strategies alone. Buprenorphine is an EBP for treating people addicted to heroin or opioid-based pain medications for non-medical use. Buprenorphine has experienced low adoption rates and is not a standard part of addiction treatment. In Ohio, the location of the study, deaths to due to accidental overdoses of opioids has increased by 304% over the past decade and surpassed auto accidents as the leading cause of accidental deaths in 2006. Ohio was selected for the study because of the public health significance of opioid abuse and because each county in Ohio acts as a stand-alone payer, offering 48 unique eligible payer environments. This trial will develop a deeper understanding of the role payers and treatment organizations play in implementing and disseminating EBPs and will focus on the public health issue of rising opioid abuse.

DETAILED DESCRIPTION:
Buprenorphine (EBP) use data will be collected from November, 2012 to May, 2016 through administrative databases located at the state of Ohio. Participants will be followed for the duration of Buprenorphine use that is an average of 5-7 months. Organizational and Payer data will be collected from January, 2013 to January, 2015. The data from the study will be analyzed and reported during January 2015 to February 2017.

ELIGIBILITY:
Inclusion Criteria:

* Treatment agencies with greater than 75 admissions per year

Exclusion Criteria:

-

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Treatment agencies and Ohio County Boards
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2016-12-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Buprenorphine Use | Five Years

CONTACTS AND LOCATIONS:
Overall Officials: Todd D Molfenter, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Ohio Department of Addiction Services, Columbus, Ohio, United States

REFERENCES:
- [Derived] Molfenter T, Kim JS, Quanbeck A, Patel-Porter T, Starr S, McCarty D. Testing use of payers to facilitate evidence-based practice adoption: protocol for a cluster-randomized trial. Implement Sci. 2013 May 10;8:50. doi: 10.1186/1748-5908-8-50. PMID 23663749